CLINICAL TRIAL: NCT04024592
Title: Reliability and Validity of Strength Measurement of the Lower Limbs in Typically Developing Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B670201834766
Record Dates: First submitted 2019-01-24; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Children; Muscle Strength; Reproducibility of Results; Muscle Strength Dynamometer; Knee
Keywords: child; dynamometry; knee joint; reproducability of results; strength testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children (Experimental)
  Interventions: Device: Biodex System 4

INTERVENTIONS:
Device: Biodex System 4 — Reliability and validity of isokinetic strength measurement of the knee, hip and ankle in typically developing children.

SUMMARY:
Reliability of isokinetic strength measurement of the knee in typically developing children has yet been studied and seems to be good. Because in daily life activities strength of the hip- and ankle-joint muscles are also important, the investigators aim to study the reliability and validity of isokinetic strength measurements of the hip and ankle.

DETAILED DESCRIPTION:
Intra-tester reliability of isokinetic strength measurements of the knee, hip and ankle in a Biodex System 4 device will be studied. Children will be assessed at different movement velocities using the test-positions as proposed by the manufacturer. Maximum peak torque will be established.

Children will also perform functional strength assessments and the relation with the results of isokinetic strength measurements will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* healthy children with good intellectual capacities

Exclusion Criteria:

* children with chronic disease or intellectual deficiency

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Isokinetic strength assessment with Biodex System 4 device | 90 minutes
  Isokinetic strength measurements of the lower limb (Max and Mean Newton Meter of 3 consecutive movements)

SECONDARY OUTCOMES:
Functional strength assessment | 30 minutes
  30 second tests (number of trials in 30 seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Van den Broeck, Professor, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided